CLINICAL TRIAL: NCT02602522
Title: The Comparison of the Effect on Danshen-Jiang-Fu Granule Prepared by Danshen (Salvia Miltiorrhiza) From Different Producing Areas (Shandong and Sichuan) for Primary Dysmenorrhea: a Cross-over, Randomized, Double-blind Controlled Trials
Brief Title: Danshen-Jiang-Fu Granule Prepared by Danshen From Different Producing Areas for Primary Dysmenorrhea
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhong Wang (Other)
Responsible Party: Sponsor-Investigator, Zhong Wang, Chief, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS-V3.0
Record Dates: First submitted 2015-11-07; First posted 2015-11-11 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Primary Dysmenorrhea; Traditional Chinese Medicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): The patients in this arm will be given 1 bag per time of Shandong Danshen-Jiang-Fu Granule, twice a day for 5 days before menorrhea and the first 2 days in the first menorrhea period. And then in the next menstrual cycle, the patients will in turn be given 1 bag per time of Sichuan Danshen-Jiang-Fu Granule, twice a day for 5 days before menorrhea and the first 2 days in the second menorrhea period.
  Interventions: Drug: Shandong Danshen-Jiang-Fu Granule; Drug: Sichuan Danshen-Jiang-Fu Granule
- controlled (Active Comparator): The patients in this arm will be given 1 bag per time of Sichuan Danshen-Jiang-Fu Granule prepared, twice a day for 5 days before menorrhea and the first 2 days in the first menorrhea period. And then in the next menstrual cycle, the patients will in turn be given 1 bag per time of Shandong Danshen-Jiang-Fu Granule, twice a day for 5 days before menorrhea and the first 2 days in the second menorrhea period.
  Interventions: Drug: Shandong Danshen-Jiang-Fu Granule; Drug: Sichuan Danshen-Jiang-Fu Granule

INTERVENTIONS:
Drug: Shandong Danshen-Jiang-Fu Granule — Danshen-Jiang-Fu Granule is prepared from 4 kinds of Chinese herbs including Danshen (Salvia Miltiorrhiza), Paojiang (Roasted Ginger), Xiangfu(Rhizoma Cyperi), Wuyao(Lindera Aggregata). The producing area of Danshen in Shandong Danshen-Jiang-Fu Granule is Laiwu District in Shandong province.
Drug: Sichuan Danshen-Jiang-Fu Granule — Danshen-Jiang-Fu Granule is prepared from 4 kinds of Chinese herbs including Danshen (Salvia Miltiorrhiza), Paojiang (Roasted Ginger), Xiangfu(Rhizoma Cyperi), Wuyao(Lindera Aggregata). The producing area of Danshen in Sichuan Danshen-Jiang-Fu Granule is Zhongjiang District in Sichuan province.

SUMMARY:
This trial aims to compare the effect of Danshen-Jiang-Fu Granule prepared by Danshen (Salvia Miltiorrhiza) from different producing areas (Shandong and Sichuan) for the relief of primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* meeting the diagnostic criteria of primary dysmenorrhea in the Primary Dysmenorrhea Consensus Guideline;
* meeting the diagnostic criteria of Hanning-xueyu(blood stasis due to cold accumulation) Zheng according to Gynecology of Chinese medicine;
* with regular menstrual cycles lasted 21 to 35 days, with menstruation lasting 3 to 9 days in the last 6 months;
* course of dysmenorrhea over 6 months;
* experienced menstrual pain scoring varying from 3cm to 6cm on a 10-cm VAS during the baseline menstrual period (one period prior to present menstrual period with treatment);
* without history of pregnancy;
* with agreement of informed consent and a working phone.

Exclusion Criteria:

* history of abdominal surgery;
* with other acute or chronic painful conditions diagnosed or suspected;
* use of hormonal contraceptives, or intra-uterine device;
* use of analgetic drugs or other analgetic treatment in the last 2 weeks;
* known allergy to Danshen (Salvia Miltiorrhiza), Paojiang (Roasted Ginger), Xiangfu(Rhizoma Cyperi) or Wuyao(Lindera Aggregata);
* prone to allergy in daily life;
* who can not complete treatment adherence to the protocol;
* attending in other trials in the last 3 months.

Ages: 14 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale on the pain of dysmenorrhea | 2 months

SECONDARY OUTCOMES:
Cox Menstrual Symptom Scale | 2 months
Daily Symptom Scale | 2 months
The change on the index of uterine artery doppler ultrasound | 2 months
  The index of uterine artery doppler ultrasound include resistance index (RI) values and the ratio between peak systolic to end-diastolic flow velocity (S/D) in uterine ascending arteries.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, Ph.D/M.D., Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences
Locations (1):
- Changzhou TCM hospital, Changzhou, Jiangsu, China